CLINICAL TRIAL: NCT05065034
Title: Effects of Antibiotic Therapy on the Short and Long-term Results of Periodontitis Treatments: Impact of Risk Factors and Treatment Characteristics
Brief Title: Effects of Antibiotic Therapy on the Short and Long-term Results of Periodontitis Treatments
Acronym: PERIODONTITIS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8333
Record Dates: First submitted 2021-09-29; First posted 2021-10-01 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Periodontitis, Adult
Keywords: Periodontitis; Inflammatory diseases; Periodontal; Teeth; Aesthetic morbidity; Cardiovascular risk; Supragingival; Subgingival; Biofilms; Prosthetic restorations
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Antibiotics are currently used in periodontology to specifically target the most pathogenic bacteria in subgingival biofilms and to improve treatments. The multiplicity of protocols / dosages tested and the variability of the results did not make it possible to reach an international consensus on antibiotic therapy and its cost / benefit ratio, in particular with regard to the significant side effects of taking antibiotics (resistance bacterial). The care environment as well as the clinical, biological and microbiological parameters can strongly influence the results in usual treatment.

ELIGIBILITY:
Inclusion criteria:

* Patient over 18 years old
* Patient treated for periodontitis between 01/01/2012 and 07/31/2021
* Patient whose medical and periodontal file contains all the elements necessary for data analysis
* Subject not having expressed, after information, his opposition to the reuse of his medical data for the purposes of this research.

Exclusion criteria:

* Patient who expressed his opposition to participating in the study
* Patient without periodontitis
* Patient smoking more than 10 cigarettes / day
* Patient presenting a dilapidated oral state (untreated caries, unrestored teeth), oral infectious foci whose management requires antibiotic treatment during the initial treatment
* Impossibility of giving the subject informed information
* Subject under safeguard of justice
* Subject under guardianship or guardianship

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient adult treated for periodontitis
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-29 (Actual); Primary Completion 2023-06-25 (Estimated); Study Completion 2023-06-25 (Estimated)

PRIMARY OUTCOMES:
A retrospective study of the use of antibiotic therapy on the short and long-term results of periodontitis treatments | Files analysed retrospectively from January 01, 2012 to July 07, 2021 will be examined]

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc DAVIDEAU, MD, PhD, Principal Investigator — Service de Médecine et de Chirurgie Bucco-Dentaires - Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Médecine et de Chirurgie Bucco-Dentaires - Hôpitaux Universitaires de Strasbourg, Strasbourg, France